CLINICAL TRIAL: NCT02442687
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Phase II Trial of JKB-121 for the Treatment of Nonalcoholic Steatohepatitis (NASH)
Brief Title: JKB-121 for the Treatment of Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manal Abdelmalek (Other)
Responsible Party: Sponsor-Investigator, Manal Abdelmalek, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00062677
Record Dates: First submitted 2015-04-07; First posted 2015-05-13 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A (Active Comparator): JKB 121, 5 mg twice daily
  Interventions: Drug: JKB-121: 5 mg twice daily
- B (Active Comparator): JKB 121, 10 mg twice daily
  Interventions: Drug: JKB-121: 10 mg twice daily
- C (Placebo Comparator): Identical appearing placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JKB-121: 5 mg twice daily
  Arms: A
Drug: JKB-121: 10 mg twice daily
  Arms: B
Drug: Placebo
  Arms: C

SUMMARY:
To evaluate the safety and potential efficacy of two dose levels of JKB-121 (5 mg twice daily and 10 mg twice daily) in reducing liver fat and/or liver biochemistry compared to placebo in patients with biopsy-proven nonalcoholic steatohepatitis

DETAILED DESCRIPTION:
JKB-121 is a long-acting small molecule that is efficacious as a weak antagonist at the TLR-4 receptor. It is a non-selective opioid antagonist which has been shown to prevent the lipopolysaccharide (LPS) induced inflammatory liver injury in a methionine/choline deficient diet fed rat model of nonalcoholic fatty liver disease. In vitro, JKB-121 neutralized or reduced the LPS-induced release of inflammatory cytokines, deactivated hepatic stellate cells, inhibited hepatic stellate cell proliferation, and collagen expression. Inhibition of the TLR4 signaling pathway may provide an effective therapy in the prevention of inflammatory hepatic injury and hepatic fibrosis in patients with nonalcoholic steatohepatitis. This study will evaluate the safety and potential efficacy of two dose levels of JKB-121 (5 mg twice daily and 10 mg twice daily) in reducing liver fat and/or liver biochemistry compared to placebo in patients with biopsy-proven nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Provision of written informed consent
3. Biopsy-proven NASH within 12 months or at screening
4. ALT > 40 U/L for women and > 60 U/L for men at screening and at least once in the previous 12 months.
5. HBA1C of ≤ 9.0

Exclusion Criteria:

1. Any chronic liver disease other than NASH
2. Cirrhosis, as assessed clinically or histologically
3. Presence of vascular liver disease
4. BMI ≤ 25 kg/m2
5. Excessive alcohol use (> 20 g/day) within the past 2 years
6. AST or ALT > 250 U/L.
7. Type 1 diabetes mellitus
8. Bariatric surgery in the past 5 years.
9. Weight gain of > 5% in past 6 months or > 10% change in past 12 months.
10. Contraindication to MRI
11. Inadequate venous access
12. HIV antibody positive, hepatitis B surface antigen positive (HBsAg), or Hepatitis C virus (HCV) RNA positive.
13. Receiving an elemental diet or parenteral nutrition
14. Chronic pancreatitis or pancreatic insufficiency
15. Any history of complications of cirrhosis
16. Concurrent conditions:

    * Inflammatory bowel disease
    * Significant cardiac disease
    * chronic infection or immune mediated disease
    * Any malignant disease
    * Prior solid organ transplant
    * Any other concurrent condition which, in the opinion of the investigator, could impact adversely on the subject participating or the interpretation of the study data.
17. Concurrent medications which may treat NASH
18. HbA1C > 9.0%
19. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2017-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manal F Abdelmalek, MD, MPH, Principal Investigator — Duke University
Locations (8):
- United States (8):
  - Digestive Disease Specialists of the Southeast, Dothan, Alabama
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Digestive Associates, Las Vegas, Nevada
  - Duke University, Durham, North Carolina
  - Digestive Disease Specialists, Cincinnati, Ohio
  - Brook Army Medical Center, Houston, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Medical College of Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027

RESULTS

PARTICIPANT FLOW:
Groups:
- JKB 5 mg BID: JKB 121, 5 mg by mouth twice daily
- JKB 10 mg BID: JKB 121, 10 mg by mouth twice daily
- Placebo BID: Identical appearing placebo by mouth twice daily
Period: Overall Study
Arm/Group | JKB 5 mg BID | JKB 10 mg BID | Placebo BID
Started | 21 | 22 | 22
Completed | 13 | 11 | 19
Not Completed | 8 | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- JKB 5 mg BID: JKB 121, 5 mg twice daily
- JKB 10 mg BID: JKB 121, 10 mg twice daily
- Placebo BID: Identical appearing placebo
- Total: Total of all reporting groups
Arm/Group | JKB 5 mg BID | JKB 10 mg BID | Placebo BID | Total
Number analyzed (Participants) | 21 | 22 | 22 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 17 | 20 | 56
  >=65 years | 2 | 5 | 2 | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 51 (11.5) | 50.5 (12.9) | 49.5 (10.5) | 51 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 17 | 44
  Male | 9 | 7 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 5 | 15
  Not Hispanic or Latino | 15 | 18 | 17 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 21 | 20 | 21 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 22 | 65
Body Mass Index [Median (Standard Deviation); unit: kg/m^2] | 40.0 (6.8) | 34.1 (6.4) | 35.4 (6.5) | 35.2 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Analysis of MRI-PDFF Change From Baseline to Week 24 (Per Protocol Population)
Time Frame: Baseline to week 24
Population: The per protocol population included only those patients with non-missing baseline (ie. screening) and the specified visit are included. If missing, the last valid measurement on or prior to the first date administration of study medication is used as baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of fat
Groups:
- JKB 121, 5 mg: JKB 121, 5 mg twice daily
  JKB-121: 5 mg twice daily
- JKB-121: 10 mg: JKB 121, 10 mg twice daily
  JKB-121: 10 mg twice daily
- Placebo: Identical appearing placebo
  Placebo
Arm/Group | JKB 121, 5 mg | JKB-121: 10 mg | Placebo
Number analyzed (Participants) | 17 | 11 | 19
percentage of fat | 0.38 [-1.95 to 2.72] | -0.44 [-3.63 to 2.74] | -3.09 [-5.28 to -0.91]
Statistical Analysis 1: Comparison: JKB 121, 5 mg vs Placebo; Test type: Other; p = 0.034, ANCOVA — The p-value was not adjusted for multiple comparison. The threshold for statistical significance was <0.05; Change from baseline as the dependent variable, baseline value as a covariate, and treatment group and diabetes stratum as factors
Statistical Analysis 2: Comparison: JKB-121: 10 mg vs Placebo; Test type: Other; p = 0.1731, ANCOVA — The p-value was not adjusted for multiple comparison. The threshold for statistical significance was <0.05; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Analysis of MRI-PDFF Change From Baseline to Week 12 (Per Protocol Population)
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Groups:
- JKB 121, 10 mg: JKB 121, 10 mg twice daily
  JKB-121: 10 mg twice daily
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 16 | 11 | 20
percentage | -1.78 [-4.05 to 0.50] | -1.50 [-4.56 to 1.56] | -2.74 [-4.78 to -0.70]
Statistical Analysis 1: Comparison: JKB 121, 5 mg vs Placebo; Test type: Other; p = 0.5276, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; The change from baseline as the dependent variable, baseline value as a covariate, and treatment group and diabetes stratum as factors
Statistical Analysis 2: Comparison: JKB 121, 10 mg vs Placebo; Test type: Other; p = 0.4968, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Analysis of ALT Change From Baseline to Week 24 (Per Protocol Population)
Time Frame: Baseline to week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 11 | 20
U/L | -6.7 [-25.2 to 11.8] | -1.3 [-25.6 to 23.0] | -20.9 [-37.7 to -4.0]
Statistical Analysis 1: Comparison: JKB 121, 5 mg vs Placebo; Test type: Other; p = 0.2591, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: JKB 121, 10 mg vs Placebo; Test type: Other; p = 0.1806, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Analysis of ALT Change From Baseline to Week 12 (Per Protocol Population)
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 11 | 20
U/L | -6.3 [-19.5 to 6.9] | -9.9 [-27.2 to 7.4] | -21.7 [-33.7 to -9.7]
Statistical Analysis 1: Comparison: JKB 121, 5 mg vs Placebo; Test type: Other; p = 0.0882, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: JKB 121, 10 mg vs Placebo; Test type: Other; p = 0.2530, ANCOVA — The p-value is not adjusted for multiple comparisons. The threshold for statistical significance was <0.05; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Remission (in Weeks)
Description: Time to remission is the time in weeks from randomization to liver function remission, defined as two consecutive ALT values within normal range (<40 U/L) during the treatment period.
Time Frame: 24 weeks
Population: No subjects reached remission; analysis not performed.
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in BMI (Body Mass Index)
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 20
kg/m^2 | -0.18 [-0.81 to 0.44] | 0.54 [-0.21 to 1.30] | -0.63 [-1.20 to -0.05]

7. Secondary Outcome: Change in Hemoglobin A1C
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1C
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 20
percentage of HbA1C | 0.07 [-0.49 to 0.63] | 0.23 [-0.44 to 0.91] | 0.45 [-0.08 to 0.98]

8. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. Optimal Range: 1.0 (0.5-1.4). Lower values represent a better outcome.
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: HOMA-IR index
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 19
HOMA-IR index | -1.013 [-3.831 to 1.805] | -0.679 [-4.132 to 2.775] | -0.404 [-3.039 to 2.231]

9. Secondary Outcome: Percent Change in Cholesterol
Time Frame: Baseline, week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 20
percent change | 6.62 [-0.42 to 13.66] | -2.55 [-11.03 to 5.94] | 2.26 [-4.18 to 8.70]

10. Secondary Outcome: Percent Change in Triglycerides
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 20
percent change | 18.12 [0.94 to 35.30] | 2.62 [-18.14 to 23.38] | 3.78 [-11.96 to 19.52]

11. Secondary Outcome: Percent Change in Low Density Lipoprotein (LDL) Cholesterol
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 18
percent change | 5.92 [-5.57 to 17.41] | -4.79 [-18.73 to 9.15] | 1.50 [-9.58 to 12.57]

12. Secondary Outcome: Percent Change in High Density Lipoprotein (HDL)
Time Frame: Baseline, week 24
Population: Only patients with non-missing baseline and the specified visit are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 20
percent change | 2.70 [-7.01 to 12.41] | -0.80 [-12.54 to 10.94] | 13.97 [5.09 to 22.86]

13. Secondary Outcome: Mean Serum Aspartate Aminotransferase (AST)
Time Frame: weeks 4, 8, 12, 16, 20, and 24
Population: Number of subjects with a result at baseline and the specified visit. Baseline is defined as the measurement at Day 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 20 | 15 | 22
U/L
  Week 4: number analyzed (Participants) | 20 | 14 | 22
  Week 4 | 45.7 (15.11) | 42.9 (12.01) | 81.0 (79.96)
  Week 8: number analyzed (Participants) | 18 | 15 | 21
  Week 8 | 45.3 (16.43) | 47.1 (15.12) | 67.4 (55.10)
  Week 12: number analyzed (Participants) | 18 | 13 | 22
  Week 12 | 47.6 (17.56) | 44.2 (16.48) | 49.7 (22.94)
  Week 16: number analyzed (Participants) | 17 | 13 | 22
  Week 16 | 42.9 (13.61) | 47.5 (22.29) | 51.1 (24.32)
  Week 20: number analyzed (Participants) | 17 | 13 | 22
  Week 20 | 50.1 (26.34) | 46.4 (27.14) | 54.0 (44.85)
  Week 24: number analyzed (Participants) | 17 | 13 | 20
  Week 24 | 49.4 (17.92) | 49.5 (33.78) | 47.4 (25.93)

14. Secondary Outcome: Mean Serum Alanine Aminotransferase (ALT)
Time Frame: weeks 4, 8, 12, 16, 20, and 24
Population: Number of subjects with a result at baseline and the specified visit. Baseline is defined as the measurement at Day 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 20 | 15 | 22
U/L
  Week 4 | 65.8 (28.28) | 70.4 (26.33) | 95.0 (66.36)
  Week 8: number analyzed (Participants) | 18 | 15 | 21
  Week 8 | 63.8 (26.03) | 77.4 (41.18) | 79.4 (42.62)
  Week 12: number analyzed (Participants) | 18 | 13 | 22
  Week 12 | 67.9 (36.23) | 65.3 (28.09) | 69.8 (39.27)
  Week 16: number analyzed (Participants) | 17 | 13 | 22
  Week 16 | 61.5 (29.06) | 69.5 (43.98) | 68.7 (33.19)
  Week 20: number analyzed (Participants) | 17 | 13 | 22
  Week 20 | 61.1 (33.08) | 63.8 (37.96) | 70.7 (43.59)
  Week 24: number analyzed (Participants) | 18 | 13 | 21
  Week 24 | 67.3 (33.80) | 68.2 (46.34) | 67.6 (48.06)

15. Secondary Outcome: Mean Serum Gamma-glutamyl Transpeptidase (GGT)
Time Frame: weeks 4, 8, 12, 16, 20, and 24
Population: Number of subjects with a result at baseline and the specified visit. Baseline is defined as the measurement at Day 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 20 | 15 | 22
U/L
  Week 4 | 68.4 (38.07) | 83.8 (48.85) | 165.0 (149.38)
  Week 8: number analyzed (Participants) | 18 | 15 | 21
  Week 8 | 73.7 (48.74) | 74.6 (35.02) | 147.5 (123.42)
  Week 12: number analyzed (Participants) | 18 | 13 | 22
  Week 12 | 79.2 (58.32) | 74.3 (36.99) | 133.8 (115.93)
  Week 16: number analyzed (Participants) | 17 | 13 | 22
  Week 16 | 78.3 (54.85) | 69.8 (33.49) | 134.7 (139.93)
  Week 20: number analyzed (Participants) | 17 | 13 | 22
  Week 20 | 75.4 (52.80) | 64.1 (30.65) | 132.9 (144.28)
  Week 24: number analyzed (Participants) | 17 | 13 | 20
  Week 24 | 86.6 (79.47) | 68.2 (30.79) | 109.7 (92.10)

16. Secondary Outcome: Number of Subjects With ALT in Normal Range at Week 24
Description: Normal range is <40 U/L
Time Frame: Week 24
Population: Number of subjects with an ALT result at the specified visit
Measure: Count of Participants; unit: Participants
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg | Placebo
Number analyzed (Participants) | 18 | 13 | 21
Participants | 5 | 4 | 7

17. Secondary Outcome: Maximum Observed Concentrations (Cmax)
Time Frame: pre-dose and at 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, and 24 hours
Population: PK Substudy Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg
Number analyzed (Participants) | 3 | 3
ng/mL | 5.26 (1.731) | 14.33 (1.986)

18. Secondary Outcome: Minimum Observed Concentration (Cmin)
Time Frame: pre-dose and at 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, and 24 hours
Population: PK Substudy Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg
Number analyzed (Participants) | 3 | 3
ng/mL | 0.349 (0.1595) | 1.512 (1.0702)

19. Secondary Outcome: Area Under Concentration-time (AUC)
Time Frame: pre-dose and at 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, and 24 hours
Population: PK Substudy Population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg
Number analyzed (Participants) | 3 | 3
h*ng/mL
  time 0 to infinity | 38.50 (13.578) | 71.24 (16.562)
  time 0 to time of last quantifiable concentration | 26.29 (9.443) | 46.55 (5.312)
  time 0 to 12 hours | 26.29 (9.443) | 50.44 (5.388)

20. Secondary Outcome: Half-life
Time Frame: pre-dose and at 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, and 24 hours
Population: PK Substudy Population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | JKB 121, 5 mg | JKB 121, 10 mg
Number analyzed (Participants) | 3 | 3
h | 8.55 (1.439) | 6.95 (2.670)

ADVERSE EVENTS:
Time Frame: 6 month
Groups:
- JKB 5 mg Twice Daily: JKB 121, 5 mg twice daily
- Placebo Twice Daily: Placebo, twice daily
- JKB 121 10 mg Twice Daily: JKB 121, 10 mg twice daily
Arm/Group | JKB 5 mg Twice Daily | Placebo Twice Daily | JKB 121 10 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 18/21 | 15/22 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JKB 5 mg Twice Daily (N=21) | Placebo Twice Daily (N=22) | JKB 121 10 mg Twice Daily (N=22)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Deemed by PI and Sponsor not be attributable to study drug
Acute on Chronic Hypoxemic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Deemed not attributable to study drub
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JKB 5 mg Twice Daily (N=21) | Placebo Twice Daily (N=22) | JKB 121 10 mg Twice Daily (N=22)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 8 (8)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Oralpharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal Congetion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Nasopharynitis (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a pilot study to assess safety and tolerability of JKB 121 in patients with biopsy-proven NASH. There The study was underpowered to detect rare events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT02442687/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT02442687/SAP_001.pdf